CLINICAL TRIAL: NCT07338656
Title: Surgery for Unstable Chest Wall Injuries - How Many Fractures Should be Fixed?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Erik Öberg Westin, Principal investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 286203
Record Dates: First submitted 2025-12-15; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Rib Fracture Multiple; Flail Chest
Keywords: Rib Fractures; Flail Chest; Traumatology; Comparative Study
MeSH Terms: conditions — Flail Chest; Rib Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization of two fractures per rib (Experimental)
  Interventions: Procedure: Surgical stabilization of two fractures per rib
- Stabilization of one fracture per rib (Active Comparator)
  Interventions: Procedure: Surgical stabilization of one fracture per rib.

INTERVENTIONS:
Procedure: Surgical stabilization of two fractures per rib — Surgical stabilization of two fractures per rib in an unstable chest wall segment.
  Arms: Stabilization of two fractures per rib
Procedure: Surgical stabilization of one fracture per rib. — Surgical stabilization of one fracture per rib in an unstable chest wall segment.
  Arms: Stabilization of one fracture per rib

SUMMARY:
The goal of this prospective, randomized study is to learn about the effects of two different surgical techniques for treating unstable chest wall injuries in adults. The main questions it aims to answer are:

Does fixing two fractures per rib lead to better healing than fixing one fracture per rib in patients with unstable chest injuries? Does the choice of surgical method affect lung function, pain, other symptoms, risk of pneumonia, or the risk of complications?

Participants will:

* Undergo surgery using either the standard method (fixing one fracture per rib) or an alternative method (fixing two fractures per rib), both using a muscle-sparing technique.
* Be followed up at 1, 3, and 12 months after surgery.
* Have CT scans at 3 months (and at 12 months if healing is incomplete) to assess bone healing.
* Be evaluated for lung function, pain, symptoms, and complications.

This study aims to provide new knowledge about which surgical method is best for unstable chest wall injuries, helping to improve treatment and recovery for these patients.

DETAILED DESCRIPTION:
Surgical treatment of chest wall injuries is an area that has attracted increased interest in the research community. It is known that rib fractures, especially unstable injuries-so-called "flail chest"-lead to pain, increased risk of pneumonia, and in some cases, the need for ventilator support and intensive care. Surgical treatment has been shown to reduce the risk of these complications. There are several described surgical methods, including large, open surgery with or without simultaneous thoracotomy, and muscle-sparing open surgery that aims to minimize damage to surrounding tissue. Thoracoscopy is used both as the main fixation method and as an adjunct to open surgery to check for intrathoracic injuries and to clear the thoracic cavity of blood. There is also a described method where a working space is created between the chest wall and the overlying tissue, and surgery is performed using thoracoscopic techniques.

There are only a few studies comparing different surgical methods. It has been shown that a muscle-sparing method resulted in shorter stays in the intensive care unit and hospital, as well as less need for ventilator support. It has also been observed that a thoracoscopic technique led to shorter hospital stays than open surgery. Muscle-sparing surgery enables stabilization of the unstable chest wall segment through one or more smaller incisions where muscle fibers are preserved during fixation. It is not clearly established how many fractures should be fixed. It has been shown that a muscle-sparing technique is advantageous compared to a method with larger incisions and thoracotomy, even if fewer ribs are fixed in the muscle-sparing method. A retrospective study from 2014 showed that the more dorsal fracture row dislocates over time if only the anterior fractures are fixed. However, it is unclear whether this has any clinical significance in the long term. We have not found any prospective study comparing fixation of both fractures in an unstable chest wall segment with fixation of only one of the fractures.

The purpose of this study is to investigate whether fixation of both fractures in an unstable chest wall segment leads to better healing than fixation of only one of the fractures. We also want to examine whether lung function improves when more fractures are fixed, whether it leads to less pain for the patient, and what symptoms related to chest wall injuries patients experience in the long term.

The project is designed as a prospective, randomized study where we compare our current muscle-sparing surgical method with fixation of only one fracture in an unstable chest wall segment with a muscle-sparing method where at least two fractures on each rib (including cartilage) in an unstable segment are fixed.

Patients are asked to participate in the study. Upon consent, patients are randomized to surgery according to clinical routine with fixation of one of the fractures on each rib in the unstable segment or surgery of two or more fractures on each rib in the unstable segment. For the unstable segment to be considered fixed, no more than two fractures on consecutive ribs may be left unfixed. Both surgical methods are performed with minimally invasive muscle-sparing technique via one or more incisions. Randomization between the two groups will be 1:1 using sealed, opaque envelopes prepared by a person independent of the study and based on a digital randomization table.

CT scans of included patients are reviewed for the presence, location, and extent of fractures on the sternum, cartilage, and ribs, as well as the presence of pneumothorax and/or hemothorax, lung contusion, and lung laceration. Injuries are graded according to AIS, presence of flail segment, ISS, and NISS. Fractures are assessed for displacement. The surgeon decides on the indication for surgery according to current guidelines (flail segment) and documents which fractures are planned to be fixed.

Demographic data collected for included patients: age, sex, height, weight, BMI, smoking status, comorbidities (COPD, asthma, pulmonary emphysema, diabetes mellitus).

The following data are collected during the hospital stay: number and length of incisions, knife time, time in hospital, time in intensive care unit and on ventilator, incidence of pneumonia, degree of pain measured with visual analogue scale (VAS), opioid equivalents, and a graphical representation on postoperative days 1, 2, and 3.

The following data are collected at follow-up visits at 1, 3, and 12 months: Radiological healing is examined with CT after 3 months. If complete radiological healing of the chest wall is lacking, a new CT is performed after 12 months. Presence of chest wall deformity and synostosis between ribs is noted. At all visits, lung function is studied with spirometry, chronic complications such as implant dysfunction and osteomyelitis, as well as pain with VAS, opioid equivalents, and a graphical representation. Patients also complete a standardized questionnaire about their symptoms.

Prospective, randomized methodological studies for fixation of rib fractures are currently lacking. It is important for method development to study the outcomes of different surgical techniques, and increased understanding of their advantages and disadvantages can greatly benefit future patients with rib fractures where surgery is indicated. The surgical technique used can affect recovery time, postoperative pain, function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery of acute (≤7 days after trauma) unstable injuries in the chest wall at the Department of Surgery, Sahlgrenska University Hospital
* Both parts of the unstable segment must be accessible for surgery.

Exclusion Criteria:

* Patients with injuries resulting from CPR
* Patients with severe head injury (Head AIS>3)
* Patients with spinal injury
* Patients with neurological or musculoskeletal disease affecting chest wall mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Radiological healing | 3 months after inclusion, 12 months after inclusion if not healed after 3 months.
  Fracture healing on CT described as "union", "non-union" or "partial union" by radiologist.

SECONDARY OUTCOMES:
Postoperative pain (opioids) | 1, 2, 3 days postoperatively and 1, 3, 12 months postoperatively.
  Pain assessed with opioid equivalents
Postoperative pain (visual analogue scale) | 1, 2, 3 days postoperatively and 1, 3, 12 months postoperatively.
  Pain assessed with a visual analogue scale.
Postoperative pain (graphical representation) | 1, 2, 3 days postoperatively and 1, 3, 12 months postoperatively.
  Pain assessed with a graphical representation of the human body where areas of pain can be indicated by the participant.
Lung function with spirometry | 1, 3 and 12 months after inclusion.
  Lung function measured with spirometry. Predicted FVC will be the outcome measure.
Complications | Up to 12 months after inclusion.
  Postoperative complications such as implant dysfunction and osteomyelitis.
Postoperative symptoms | 1, 3 and 12 months after inclusion.
  Standardized questionnaire regarding postoperative symptoms such as tightness, shortness of breath.
Time in hospital | From inclusion and up to 12 months after.
  Time spent in hospital after initial trauma
Time in intensive care unit | From inclusion and up to 12 months after.
  Time in intensive care unit after initial trauma.
Time in ventilator | From inclusion and up to 12 months after.
  Time in ventilator after initial trauma.
Incidence of pneumonia | Up to 30 days after inclusion.
  Incidence of pneumonia defined as radiological imaging consistent with pneumonia combined with typical symptoms (cough, shortness of breath, fever) or positive sputum culture.

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Corina Caragounis, Ph.D, Ass. Prof, Study Director — Institution of Clinical Sciences, Sahlgrenska Academy, Gothenburg University. Department of Surgery, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sermonesi G, Bertelli R, Pieracci FM, Balogh ZJ, Coimbra R, Galante JM, Hecker A, Weber D, Bauman ZM, Kartiko S, Patel B, Whitbeck SS, White TW, Harrell KN, Perrina D, Rampini A, Tian B, Amico F, Beka SG, Bonavina L, Ceresoli M, Cobianchi L, Coccolini F, Cui Y, Dal Mas F, De Simone B, Di Carlo I, Di Saverio S, Dogjani A, Fette A, Fraga GP, Gomes CA, Khan JS, Kirkpatrick AW, Kruger VF, Leppaniemi A, Litvin A, Mingoli A, Navarro DC, Passera E, Pisano M, Podda M, Russo E, Sakakushev B, Santonastaso D, Sartelli M, Shelat VG, Tan E, Wani I, Abu-Zidan FM, Biffl WL, Civil I, Latifi R, Marzi I, Picetti E, Pikoulis M, Agnoletti V, Bravi F, Vallicelli C, Ansaloni L, Moore EE, Catena F. Surgical stabilization of rib fractures (SSRF): the WSES and CWIS position paper. World J Emerg Surg. 2024 Oct 18;19(1):33. doi: 10.1186/s13017-024-00559-2. PMID 39425134
- [Background] Marasco S, Liew S, Edwards E, Varma D, Summerhayes R. Analysis of bone healing in flail chest injury: do we need to fix both fractures per rib? J Trauma Acute Care Surg. 2014 Sep;77(3):452-8. doi: 10.1097/TA.0000000000000375. PMID 25159250
- [Background] Tichenor M, Reparaz LB, Watson C, Reeves J, Prest P, Fitzgerald M, Patel N, Tan X, Hessey J. Intrathoracic plates versus extrathoracic plates: a comparison of postoperative pain in surgical stabilization of rib fracture technique. Trauma Surg Acute Care Open. 2023 Nov 3;8(1):e001201. doi: 10.1136/tsaco-2023-001201. eCollection 2023. PMID 37936903
- [Background] Tay-Lasso E, Alaniz L, Grant W, Hovis G, Frank M, Kincaid C, Brynn S, Pieracci FM, Nahmias J, Barrios C, Rockne W, Chin T, Swentek L, Schubl SD. Prospective single-center paradigm shift of surgical stabilization of rib fractures with decreased length of stay and operative time with an intrathoracic approach. J Trauma Acute Care Surg. 2023 Apr 1;94(4):567-572. doi: 10.1097/TA.0000000000003811. Epub 2022 Oct 25. PMID 36301075
- [Background] Oberg Westin E, Fagevik Olsen M, Ortenwall P, Caragounis EC. Retrospective comparison of operative technique for chest wall injuries. Injury. 2023 Mar 10:S0020-1383(23)00248-6. doi: 10.1016/j.injury.2023.03.012. Online ahead of print. PMID 36925375
- [Background] Xia H, Zhu P, Li J, Zhu D, Sun Z, Deng L, Zhang Y, Wang D. Thoracoscope combined with internal support system of chest wall in open reduction and internal fixation for multiple rib fractures. Exp Ther Med. 2018 Dec;16(6):4650-4654. doi: 10.3892/etm.2018.6817. Epub 2018 Oct 1. PMID 30542416
- [Background] Fraser SF, Tan C, Kuppusamy MK, Gukop P, Hunt IJ. The role of a video-assisted thoracic approach for rib fixation. Eur J Trauma Emerg Surg. 2017 Apr;43(2):185-190. doi: 10.1007/s00068-016-0641-1. Epub 2016 Feb 5. PMID 26850079
- [Background] Nowack T, Nonnemacher C, Christie DB. Video-Assisted Thoracoscopic Surgery as an Adjunct to Rib Fixation. Am Surg. 2022 Jun;88(6):1338-1340. doi: 10.1177/0003134820943642. Epub 2020 Aug 26. No abstract available. PMID 32845731
- [Background] Zhang J, Hong Q, Mo X, Ma C. Complete Video-assisted Thoracoscopic Surgery for Rib Fractures: Series of 35 Cases. Ann Thorac Surg. 2022 Feb;113(2):452-458. doi: 10.1016/j.athoracsur.2021.01.065. Epub 2021 Mar 3. PMID 33675706
- [Background] Pieracci FM, Johnson JL, Stovall RT, Jurkovich GJ. Completely thoracoscopic, intra-pleural reduction and fixation of severe rib fractures. Trauma Case Rep. 2015 Nov 4;1(5-8):39-43. doi: 10.1016/j.tcr.2015.10.001. eCollection 2015 Oct. No abstract available. PMID 30101174
- [Background] Bauman ZM, Beard R, Cemaj S. When less is more: A minimally invasive, intrathoracic approach to surgical stabilization of rib fractures. Trauma Case Rep. 2021 Mar 11;32:100452. doi: 10.1016/j.tcr.2021.100452. eCollection 2021 Apr. PMID 33778146
- [Background] Schulz-Drost S, Grupp S, Pachowsky M, Oppel P, Krinner S, Mauerer A, Hennig FF, Langenbach A. Stabilization of flail chest injuries: minimized approach techniques to treat the core of instability. Eur J Trauma Emerg Surg. 2017 Apr;43(2):169-178. doi: 10.1007/s00068-016-0664-7. Epub 2016 Mar 22. PMID 27084543
- [Background] Marasco S, Saxena P. Surgical rib fixation - technical aspects. Injury. 2015 May;46(5):929-32. doi: 10.1016/j.injury.2014.12.021. Epub 2015 Jan 10. PMID 25624272
- [Background] Gasparri MG, Tisol WB, Haasler GB. Rib stabilization: lessons learned. Eur J Trauma Emerg Surg. 2010 Oct;36(5):435-40. doi: 10.1007/s00068-010-0048-3. Epub 2010 Sep 24. PMID 26816224
- [Background] Granhed HP, Pazooki D. A feasibility study of 60 consecutive patients operated for unstable thoracic cage. J Trauma Manag Outcomes. 2014 Dec 30;8(1):20. doi: 10.1186/s13032-014-0020-z. eCollection 2014. PMID 25642282
- [Background] Bottlang M, Long WB, Phelan D, Fielder D, Madey SM. Surgical stabilization of flail chest injuries with MatrixRIB implants: a prospective observational study. Injury. 2013 Feb;44(2):232-8. doi: 10.1016/j.injury.2012.08.011. Epub 2012 Aug 19. PMID 22910817
- [Background] Liu T, Liu P, Chen J, Xie J, Yang F, Liao Y. A Randomized Controlled Trial of Surgical Rib Fixation in Polytrauma Patients With Flail Chest. J Surg Res. 2019 Oct;242:223-230. doi: 10.1016/j.jss.2019.04.005. Epub 2019 May 14. PMID 31100568
- [Background] Marasco SF, Davies AR, Cooper J, Varma D, Bennett V, Nevill R, Lee G, Bailey M, Fitzgerald M. Prospective randomized controlled trial of operative rib fixation in traumatic flail chest. J Am Coll Surg. 2013 May;216(5):924-32. doi: 10.1016/j.jamcollsurg.2012.12.024. Epub 2013 Feb 13. PMID 23415550
- [Background] Granetzny A, Abd El-Aal M, Emam E, Shalaby A, Boseila A. Surgical versus conservative treatment of flail chest. Evaluation of the pulmonary status. Interact Cardiovasc Thorac Surg. 2005 Dec;4(6):583-7. doi: 10.1510/icvts.2005.111807. Epub 2005 Sep 15. PMID 17670487
- [Background] Tanaka H, Yukioka T, Yamaguti Y, Shimizu S, Goto H, Matsuda H, Shimazaki S. Surgical stabilization of internal pneumatic stabilization? A prospective randomized study of management of severe flail chest patients. J Trauma. 2002 Apr;52(4):727-32; discussion 732. doi: 10.1097/00005373-200204000-00020. PMID 11956391
- [Background] Ciraulo DL, Elliott D, Mitchell KA, Rodriguez A. Flail chest as a marker for significant injuries. J Am Coll Surg. 1994 May;178(5):466-70. PMID 8167883
- [Background] Sirmali M, Turut H, Topcu S, Gulhan E, Yazici U, Kaya S, Tastepe I. A comprehensive analysis of traumatic rib fractures: morbidity, mortality and management. Eur J Cardiothorac Surg. 2003 Jul;24(1):133-8. doi: 10.1016/s1010-7940(03)00256-2. PMID 12853057
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614